CLINICAL TRIAL: NCT03385304
Title: Aqueous-PREP: A Pragmatic Randomized Trial Evaluating Pre-operative Aqueous Antiseptic Skin Solutions in Open Fractures
Brief Title: Pre-operative Aqueous Antiseptic Skin Solutions in Open Fractures
Acronym: Aqueous-PREP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: McMaster University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gerard Slobogean, Assistant Professor, Department of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00078470
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Surgical Site Infection; Unplanned Fracture-Related Reoperation; Open Appendicular Fracture
Keywords: Surgical Site Infection; Open Fracture; Povidone-iodine; Chlorhexidine gluconate; Peri-operative Preparation Solutions
MeSH Terms: conditions — Surgical Wound Infection; Fractures, Open | interventions — Povidone-Iodine; chlorhexidine gluconate; Chromogranins

STUDY DESIGN:
Intervention Model Description: Treatment allocation will be determined using a cluster-randomized crossover trial design. The order of treatment allocation for each orthopaedic practice will be randomly assigned using a computer generated randomization table. Each site will start with the initially allocated study solution and eventually crossover to the other solution for their second recruitment period. This process of alternating treatments will repeat approximately every 2 months as dictated by the initial randomization.
Who Masked: Outcomes Assessor
Masking Description: The orthopaedic team (including the study coordinators) cannot be blinded to the treatment allocation as the antiseptic solutions are visually distinguishable and these individuals need to lead the implementation of the cluster-crossover protocol at their clinical site. The Adjudication Committee Members and data analysts will be blinded to the study treatment. All interpretation of study results will initially be done in a blinded manner by developing two interpretations of the results. One interpretation will assume treatment A is povidone-iodine, the other interpretation will assume it is CHG. Once the data interpretations for each assumption are finalized, the data will be unblinded and the correct interpretation will be accepted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 10% povidone-iodine (1% free iodine) in purified water (Experimental): The povidone-iodine solution will contain 10% povidone-iodine (1% free iodine) in purified water as the only active ingredient. Operating room personnel will apply the solution to the operative site as the final preoperative skin antisepsis preparation immediately prior to commencing surgical fixation. They will apply the solution as per manufacturer's directions for use (e.g., technique of application, duration of application, drying time, drying techniques, replacement of draping, etc.).
  Interventions: Drug: 10% povidone-iodine (1% free iodine) in purified water; Drug: 4% chlorhexidine gluconate (CHG) in purified water
- 4% chlorhexidine gluconate (CHG) in purified water (Experimental): The CHG solution will contain 4% CHG in purified water as the only active ingredient. Operating room personnel will apply the solution to the operative site as the final preoperative skin antisepsis preparation immediately prior to commencing surgical fixation. They will apply the solution as per manufacturer's directions (e.g., technique of application, duration of application, drying time, replacement of draping, etc.).
  Interventions: Drug: 10% povidone-iodine (1% free iodine) in purified water; Drug: 4% chlorhexidine gluconate (CHG) in purified water

INTERVENTIONS:
Drug: 10% povidone-iodine (1% free iodine) in purified water — Participant recruitment will begin with the clinical sites using their assigned pre-operative antiseptic skin solution for all open fracture surgeries for a two-month period.
Drug: 4% chlorhexidine gluconate (CHG) in purified water — Once the first intervention phase is completed, each site will crossover to the opposite study solution. Each site will need to develop local procedures to ensure a successful crossover. They will use the second solution for all open fracture surgeries for a two-month period, and will then crossover back to the solution in the first intervention phase.

SUMMARY:
The prevention of infection is the single most important goal influencing peri-operative care of patients with open fractures. Standard practice in the management of open fractures includes sterile technique and pre-operative skin preparation with an antiseptic solution. The available solutions kill bacteria and decrease the quantity of native skin flora, thereby decreasing surgical site infection (SSI). While there is extensive guidance on specific procedures for prophylactic antibiotic use and standards for sterile technique, the evidence regarding the choice of antiseptic skin preparation solution is very limited for open fracture surgery.

ELIGIBILITY:
The inclusion criteria are:

1. Patients 18 years of age or older.
2. Open fracture of the appendicular skeleton.
3. Received or will receive definitive fracture treatment with a surgical implant(s) (e.g., internal fixation, external fixation, joint prosthesis, etc.).
4. Open fracture wound management that includes formal surgical debridement within 72 hours of their injury.
5. Will have all planned fracture care surgeries performed by a participating surgeon or delegate.
6. Informed consent obtained.
7. Patient enrolled within 3 weeks of their fracture.

The exclusion criteria are:

1. Patients that did not or will not receive the allocated pre-operative surgical preparation solution due to a medical contraindication.
2. Received previous surgical debridement or management of their open fracture at a non-participating hospital or clinic.
3. Open fracture managed outside of the participating orthopaedic service (e.g., hand fracture managed by plastic surgeon).
4. Chronic or acute infection at or near the fracture site at the time of initial fracture surgery.
5. Burns at the fracture site.
6. Incarceration.
7. Expected injury survival of less than 90 days.
8. Terminal illness with expected survival less than 90 days.
9. Previous enrollment in a PREP-IT trial.
10. Currently enrolled in a study that does not permit co-enrollment.
11. Unable to obtain informed consent due to language barriers.
12. Likely problems, in the judgment of study personnel, with maintaining follow-up with the patient.
13. Excluded due to sampling strategy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1638 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Slobogean, MD, Principal Investigator — University of Maryland, Baltimore; Sheila Sprague, PhD, Principal Investigator — McMaster University; Mohit Bhandari, MD, Principal Investigator — McMaster University
Locations (15):
- United States (11):
  - The CORE Institute / Banner University Medical Center, Phoenix, Arizona
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Wright State University / Miami Valley Hospital, Dayton, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - McGovern Medical School at University of Texas Health Science Center Houston, Houston, Texas
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - McMaster University, Center for Evidence-Based Orthopaedics, Hamilton, Ontario
- Spain (2):
  - Hospital Parc Tauli de Sabadell, Barcelona
  - Vall d'Hebron University Hospital, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Hara NN, Heels-Ansdell D, Bzovsky S, Dodds S, Thabane L, Bhandari M, Guyatt G, Devereaux PJ, Slobogean GP, Sprague S; PREP-IT Investigators. A pragmatic randomized trial evaluating pre-operative aqueous antiseptic skin solutions in open fractures (Aqueous-PREP): statistical analysis plan. Trials. 2022 Sep 12;23(1):772. doi: 10.1186/s13063-022-06541-0. PMID 36096826
- [Derived] PREP-IT Investigators. Aqueous skin antisepsis before surgical fixation of open fractures (Aqueous-PREP): a multiple-period, cluster-randomised, crossover trial. Lancet. 2022 Oct 15;400(10360):1334-1344. doi: 10.1016/S0140-6736(22)01652-X. PMID 36244384
- [Derived] Sprague S, Guyatt P, Bzovsky S, Nguyen U, Bhandari M, Thabane L, Petrisor B, Johal HS, Leonard J, Dodds S, Mossuto F, O'Toole RV, Howe A, Demyanovich HK, Camara M, O'Hara NN, Slobogean GP; PREP-IT Investigators. Pragmatic randomized trial evaluating pre-operative aqueous antiseptic skin solution in open fractures (Aqueous-PREP): the feasibility of a cluster randomized crossover study. Pilot Feasibility Stud. 2021 Mar 1;7(1):61. doi: 10.1186/s40814-021-00800-8. PMID 33648577
- [Derived] Sprague S, Scott T, Dodds S, Pogorzelski D, McKay P, Harris AD, Wood A, Thabane L, Bhandari M, Mehta S, Gaski G, Boulton C, Marcano-Fernandez F, Guerra-Farfan E, Hebden J, O'Hara LM, Slobogean GP; PREP-IT Investigators. Cluster identification, selection, and description in cluster randomized crossover trials: the PREP-IT trials. Trials. 2020 Aug 12;21(1):712. doi: 10.1186/s13063-020-04611-9. PMID 32787892
- [Derived] Program of Randomized Trials to Evaluate Pre-operative Antiseptic Skin Solutions in Orthopaedic Trauma (PREP-IT) Investigators; Slobogean GP, Sprague S, Wells J, Bhandari M, Rojas A, Garibaldi A, Wood A, Howe A, Harris AD, Petrisor BA, Mullins DC, Pogorzelski D, Marvel D, Heels-Ansdell D, Mossuto F, Grissom F, Del Fabbro G, Guyatt GH, Della Rocca GJ, Demyanovich HK, Gitajn IL, Palmer J, D'Alleyrand JC, Friedrich J, Rivera J, Hebden J, Rudnicki J, Fowler J, Jeray KJ, Thabane L, Marchand L, O'Hara LM, Joshi MG, Talbot M, Camara M, Szasz OP, O'Hara NN, McKay P, Devereaux PJ, O'Toole RV, Zura R, Morshed S, Dodds S, Li S, Tanner SL, Scott T, Nguyen U. Effectiveness of Iodophor vs Chlorhexidine Solutions for Surgical Site Infections and Unplanned Reoperations for Patients Who Underwent Fracture Repair: The PREP-IT Master Protocol. JAMA Netw Open. 2020 Apr 1;3(4):e202215. doi: 10.1001/jamanetworkopen.2020.2215. PMID 32259266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 8, 2018, and June 8, 2021 at 14 hospitals in Canada, Spain and the USA. Eligible patients were adults aged 18 years or older with an open extremity fracture treated with a surgical fixation implant. For inclusion, the open fracture required formal surgical debridement within 72 hours of the injury.
Pre-assignment Details: To ensure wide generalizability to routine practice, the protocol allowed prewashing of the operative extremity with alcohol or other antiseptics before performing the final skin antisepsis with the study solution. In addition to ensuring trial feasibility and protocol adherence, this decision pragmatically allowed the intact skin to receive mechanical scrubbing or partial alcohol antisepsis at the treating surgeon's discretion.
Units Other Than Participants: Clinical Sites
Period: Overall Study
Arm/Group | 10% Povidone-iodine (1% Free Iodine) in Purified Water | 4% Chlorhexidine Gluconate (CHG) in Purified Water
Started (Total Study Duration) | 828; 7 Clinical Sites | 810; 7 Clinical Sites
Months 1-2 | 114; 7 Clinical Sites | 108; 7 Clinical Sites
Months 3-4 | 102; 7 Clinical Sites | 104; 7 Clinical Sites
Months 5-6 | 98; 7 Clinical Sites | 53; 5 Clinical Sites
Months 7-8 | 50; 5 Clinical Sites | 68; 7 Clinical Sites
Months 9-10 | 91; 6 Clinical Sites | 63; 5 Clinical Sites
Months 11-12 | 72; 5 Clinical Sites | 75; 5 Clinical Sites
Months 13-14 | 62; 5 Clinical Sites | 50; 4 Clinical Sites
Months 15-16 | 38; 4 Clinical Sites | 55; 5 Clinical Sites
Months 17-18 | 38; 5 Clinical Sites | 44; 5 Clinical Sites
Months 19-20 | 32; 5 Clinical Sites | 46; 3 Clinical Sites
Months 21-22 | 50; 4 Clinical Sites | 40; 5 Clinical Sites
Months 23-24 | 30; 4 Clinical Sites | 64; 5 Clinical Sites
Months 25-26 | 22; 1 Clinical Sites | 14; 1 Clinical Sites
Months 27-28 | 21; 1 Clinical Sites | 18; 1 Clinical Sites
Months 29-30 | 0; 0 Clinical Sites | 8; 1 Clinical Sites
Months 31-32 | 8; 1 Clinical Sites | 0; 0 Clinical Sites
Completed (Total Study Duration) | 787; 7 Clinical Sites | 784; 7 Clinical Sites
Not Completed | 41; 0 Clinical Sites | 26; 0 Clinical Sites
Not completed — Death | 19 | 7
Not completed — Lost to Follow-up | 17 | 14
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Incarceration | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10% Povidone-iodine (1% Free Iodine) in Purified Water | 4% Chlorhexidine Gluconate (CHG) in Purified Water | Total
Number analyzed (Participants) | 828 | 810 | 1638
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 45.2 (18.2) | 44.5 (17.9) | 44.9 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 324 | 303 | 627
  Male | 504 | 507 | 1011
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 665 | 624 | 1289
  Race: Black | 124 | 137 | 261
  Race: Central or South American | 10 | 20 | 30
  Race: Asian | 8 | 10 | 18
  Race: Prefer not to answer | 7 | 11 | 18
  Race: Indigenous | 11 | 5 | 16
  Race: Multiracial | 3 | 2 | 5
  Race: Native Hawaiian or Pacific Islander | 0 | 1 | 1
BMI [Count of Participants; unit: Participants] — BMI (Body Mass Index) [kg/m^2] was determined by collecting each participant's weight and height
  Participants
    Underweight (<18.5 kg/m^2) | 9 | 10 | 19
    Healthy weight (18.5 - 24.9 kg/m^2) | 243 | 200 | 443
    Overweight (25.0-29.9 kg/m^2) | 247 | 271 | 518
    Obesity (>30.0 kg/m^2) | 329 | 329 | 658
Diabetes of any type [Count of Participants; unit: Participants] | 94 | 76 | 170
Current smoker [Count of Participants; unit: Participants] | 293 | 274 | 567
American Society of Anesthesiologist (ASA) Physical Score [Count of Participants; unit: Participants] — The American Society of Anesthesiologist (ASA) score is a subjective assessment of a patient's overall health that is based on five classes (I to V).
  I. Patient is a completely healthy fit patient. II. Patient has mild systemic disease. III. Patient has severe systemic disease that is not incapacitating. IV. Patient has incapacitating disease that is a constant threat to life. V. A moribund patient who is not expected to live 24 hour with or without surgery.
  Participants
    Class I or II | 423 | 436 | 859
    Class III or higher | 405 | 374 | 779
Number of included open fractures per participant [Count of Participants; unit: Participants]
  One | 775 | 753 | 1528
  Two | 44 | 51 | 95
  Three | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Superficial Incisional Surgical Site Infection (SSI)
Description: Guided by the Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network reporting criteria (2017):
  Date of event for infection may occur from the date of fracture to 30 days after the definitive fracture management surgery; AND involves only skin and subcutaneous tissue of the incision; AND patient has at least one of the following:
  1. purulent drainage from the superficial incision.
  2. organisms identified from an aseptically obtained specimen from the superficial incision or subcutaneous tissue by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment
  3. superficial incision that is deliberately opened by a surgeon, and culture or non-culture-based testing is not performed. AND patient has at least one of the following signs or symptoms: pain or tenderness; localized swelling; erythema; or heat.
  4. diagnosis of a superficial incisional SSI by the surgeon.
Time Frame: Within 30 days of the patient's last planned fracture management surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 10% Povidone-iodine (1% Free Iodine) in Purified Water | 4% Chlorhexidine Gluconate (CHG) in Purified Water
Number analyzed (Participants) | 787 | 784
Participants | 13 | 7

2. Primary Outcome: Number of Participants With a Deep Incisional or Organ/Space Infection
Description: Guided by CDC's National Healthcare Safety Network Surgical Site Infection reporting criteria (2017):
  Deep Incisional Infection:
  Occurs within 90 days post definitive fracture management; & involves fascial/muscle layers; & has at least one of the following:
  1. deep incision purulent drainage
  2. a deep incision that dehisces, or is opened by a surgeon, and organism is identified by microbiologic testing; or microbiologic testing is not performed & has at least one of the following: fever (> 38 °C); localized pain or tenderness
  3. other evidence of deep incision infection on anatomical exam or imaging test
  Organ/Space Infection:
  Occurs within 90 days post definitive fracture management; & involves any part of the body deeper than the fascial/muscle layers; & has at least one of the following:
  1. organ/space purulent drainage
  2. organisms in organ/space identified by microbiologic testing
  3. other evidence of organ/space infection on anatomical exam or imaging test
Time Frame: Within 90 days of the patient's last planned fracture management surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 10% Povidone-iodine (1% Free Iodine) in Purified Water | 4% Chlorhexidine Gluconate (CHG) in Purified Water
Number analyzed (Participants) | 787 | 784
Participants | 46 | 51

3. Secondary Outcome: Number of Participants With an Unplanned Fracture-Related Reoperation
Description: Common examples include any unplanned fracture-related surgery that is associated with an infection at the operative site or contiguous to it, a wound-healing problem, or a fracture delayed union or non-union.
Time Frame: Within 12 months of the patient's last planned operation
Population: Primary and secondary outcomes were evaluated using a complete case analysis. For that reason, the overall number of participants analyzed differs from the numbers provided under the Participant Flow module.
Measure: Count of Participants; unit: Participants
Arm/Group | 10% Povidone-iodine (1% Free Iodine) in Purified Water | 4% Chlorhexidine Gluconate (CHG) in Purified Water
Number analyzed (Participants) | 734 | 738
Participants | 118 | 115

ADVERSE EVENTS:
Time Frame: 1 year post injury
Description: This study did not collect data regarding "Other (Not Including Serious) Adverse Events".
Arm/Group | 10% Povidone-iodine (1% Free Iodine) in Purified Water | 4% Chlorhexidine Gluconate (CHG) in Purified Water
All-Cause Mortality (participants affected / at risk) | 19/828 | 7/810
Serious Adverse Events (participants affected / at risk) | 365/828 | 368/810
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10% Povidone-iodine (1% Free Iodine) in Purified Water (N=828) | 4% Chlorhexidine Gluconate (CHG) in Purified Water (N=810)
Study Fracture Related Complication (Musculoskeletal and connective tissue disorders) | 178 (178) | 192 (192)
Non-Study Fracture Related Complication (Musculoskeletal and connective tissue disorders) | 23 (23) | 31 (31)
Neurological (Nervous system disorders) | 5 (5) | 8 (8)
Renal (Renal and urinary disorders) | 10 (10) | 10 (10)
Cardiac (Cardiac disorders) | 7 (7) | 9 (9)
Vascular (Vascular disorders) | 11 (11) | 12 (12)
Gastro-Intestinal (Gastrointestinal disorders) | 10 (10) | 12 (12)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 25 (25)
Other (General disorders) | 95 (95) | 69 (69)

LIMITATIONS AND CAVEATS:
The uncontrolled use of adjunctive skin preparations before final antisepsis is a potential limitation of our study design. Although the use of a prewash with adjunctive alcohol was similarly distributed between the treatment groups, post-randomization confounding from this practice might exist. The trial has other limitations, including unmasked treatment allocation and the decision to initiate each recruitment site as soon as possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT03385304/Prot_SAP_000.pdf